CLINICAL TRIAL: NCT03636594
Title: "Let's Boogie": Feasibility of a Dance Intervention in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Feasibility of Dance in People With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Principal Investigator, Roger Goldstein, Clinical Professor, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-023-WP
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: COPD
Keywords: Dance; COPD; Maintenance program; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance (Experimental): This was a single arm study with all participants receiving the same intervention.
  Interventions: Other: Dance

INTERVENTIONS:
Other: Dance — The dance program consisted of one-hour dance classes delivered twice a week for 8 weeks. The classes featured different dance types (such as partnered and non-partnered) and genres (such as salsa, ballroom and jazz) with increasing complexity.

SUMMARY:
Despite the benefits associated with individuals with chronic obstructive pulmonary disease (COPD) engaging in pulmonary rehabilitation (PR) programs, the benefits diminish by 6 months. A new innovative approach is needed to increase motivation to exercise and to minimize diminution of effect. Dance is a fun and interactive activity, which has shown benefits in other populations, such as Parkinson's disease and stroke. The aim of this study was to investigate the feasibility of dance in individuals with COPD following PR.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by spirometry (FEV1/FVC < 0.7)
* Adequate communication with or without corrective hearing aids
* No intensive PR for at least 6 months before recruitment
* An ability to provide informed consent.

Exclusion Criteria:

* Presence of comorbidities that could have prevented communication or safe exercise

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 8 weeks
  Enrollment rate is calculated as a percentage (number of people enrolled/ number of people approached)
Attendance rate | 8 weeks
  Attendance rate is calculated as a mean percentage for the group (number of sessions attended/ number of total sessions)
Participant satisfaction and perceived benefits (Participant satisfaction questionnaire) questionnaire | 8 weeks
  Participant satisfaction and the perceived benefits were assessed by asking participants to complete a nine-item survey which asked participants to report their level of agreement with statements on enjoyment and perceived improvements or benefits according to a 5-point Likert type scale (1 = strongly agree, 5 = strongly disagree). The questionnaire contained open-ended questions asking participants what they liked best and least as well as what they would change about the intervention.
Occurrence of adverse events | 8 weeks
  Adverse events were tracked and the program is considered safe and feasible if no adverse events occurred.

SECONDARY OUTCOMES:
Change in functional capacity (6-minute walk test) | Change from baseline to end of 8-week dance program
  Changes in the distance walked as measured using 6-minute walk test. The farther the distance walked in 6 minutes, the better the functional capacity.
Change in Balance Evaluation Systems Test (BESTest) score | Change from baseline to end of 8-week dance program
  Change in balance from baseline to end of 8-week dance program as measured by Balance Evaluation Systems Test (BESTest). The BESTest consists of 36 items that evaluate balance impairments across six postural control contexts. These six contexts are: biomechanical constraints, stability limits/verticality, anticipatory postural adjustments, postural responses, sensory orientation and stability in gait. Total score of BESTest is 108 points (the item-level score ranges from 0 "severe impairment to 3 "no impairment"), calculated into a percentage score (0%-100%) with the higher score the better the balance.
Change in Berg Balance Scale score | Change from baseline to end of 8-week dance program
  Change in balance from baseline to end of 8-week dance program as measured by Balance Evaluation Systems Test (BESTest) and Berg balance scale. Berg balance scale comprises a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores, with a higher score indicating better balance.
Change in balance confidence (activities specific balance scale) | Change from baseline to end of 8-week dance program
  Change in balance confidence from baseline to end of 8-week dance program as measured using the Activities-specific Balance Confidence (ABC) scale. The scale consists of 16 statements on different activities and the participant indicates their level of confidence in doing the activities without losing their balance or becoming unsteady from choosing one of the percentage points on the scale from 0% to 100% with the higher values represent a better balance confidence.
Change in anxiety and depression (hospital anxiety and depression scale) | Change from baseline to end of 8-week dance program
  Change in anxiety and depression from baseline to end of 8-week dance program measured using Hospital Anxiety and Depression Scale.The scale consisted of 14 items (seven for anxiety and the same for depression). Each item is a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression with the lower score is the better outcome
Change in health related quality of life (chronic respiratory disease questionnaire) | Change from baseline to end of 8-week dance program
  Change in health related quality of life from baseline to end of 8-week dance program measured using the chronic respiratory questionnaire which is an interviewer-administered one that measures both physical and emotional aspects of chronic respiratory disease. The questionnaire is a 7-point modified Likert Scale, consists of 20 items that explore four categories: dyspnea, fatigue, emotional function and mastery. The maximum score possible is 140 and the lowest is 20 with the higher scores indicate better health-related quality of life
Change in step count | Change from baseline to end of 8-week dance program
  Measured using Fitbit charge2 physical activity trackers.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Study Chair — University of Toronto
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available upon request and up to 7 years after publication